CLINICAL TRIAL: NCT01076322
Title: A Study to Evaluate the Efficacy and Safety of Meptin® Swinghaler® and Ventolin® MDI in Stable Asthma Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Taiwan Otsuka Pharm. Co., Ltd (Industry)
Responsible Party: Edward C.Y. Peng, Taiwan Otsuka Pharmaceutical Co., Ltd
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 002-TWB-0801
Record Dates: First submitted 2010-02-24; First posted 2010-02-26 (Estimated); Last update posted 2010-08-12 (Estimated); Status verified 2010-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Albuterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment-A sequence (Experimental): Meptin® Swinghaler / Ventolin® MDI
  Interventions: Drug: Meptin® Swinghaler; Drug: Ventolin® MDI
- Treatment-B sequence (Experimental): Ventolin® MDI / Meptin® Swinghaler
  Interventions: Drug: Meptin® Swinghaler; Drug: Ventolin® MDI

INTERVENTIONS:
Drug: Meptin® Swinghaler — Meptin® Swinghaler®
  * Ingredient: Procaterol HCL
  * Dosage form: 10g/puff
  * Dose(s): 10g
  * Dosing schedule: 20g (total 20g)
  Other Names: Meptin® Swinghaler®; Procaterol HCL; Ventolin® MDI; Salbutamol sulfate
Drug: Ventolin® MDI — Ventolin® MDI
  * Ingredient: Salbutamol sulfate
  * Dosage form: 100g/puff
  * Dose(s): 100g
  * Dosing schedule: 200g (total 200g)

SUMMARY:
This is an open-label, randomized, cross-over, active-controlled study to evaluate the efficacy and safety effects using Meptin® Swinghaler and Ventolin® MDI in stable asthma patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male or females outpatients aged ≥ 16 years old with stable mild to moderate persistent asthma; Stability was assessed the patient remained in the same severity class (mild, moderate) and had no acute exacerbations by investigator judgment during the past 14 days;
2. Pulmonary function test:

   * Improvement ≥12% reversibility in FEV1 or FVC following administration of an inhaled β2-agonist before the study or ;
   * Positive result of Broncho-provocation test (PC20 ≤ 32 mg/ml) before the study.
3. Baseline forced expiratory volume in one second 60% ≤(FEV1)≤ 90% of predicted value on entry of the study;

Exclusion Criteria:

1. Hypersensitivity to β2-agonist or lactose;
2. Hospitalization due to asthma during the previous 3months;
3. Respiratory tract infection requiring treatment with antibiotics in the previous 4 weeks;
4. Oral or systemic corticosteroids in the previous 4weeks;
5. Inadequately controlled hyperthyroidism;
6. Severe hepatic or renal or cardiovascular disease as judged by the investigator;
7. Patients receive an investigational drug within 30 days prior to admission to the study;
8. Patients with significant alcohol, drug or medication abuse as judged by the investigator;
9. Females who are pregnant or breast-feeding; (exception: Females of child-bearing age might be included, if in the opinion of the investigator, they are using adequate contraceptive precautions).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
The change in Forced Expiratory Volume in 1 second (FEV1) value. | 2 days

SECONDARY OUTCOMES:
The change in sGaw | 2 days
The changes in IOS parameters (R, X and RF) | 2 days
The change in Peak Expiratory Flow Rate (PEFR) | 2 days
The change in Forced Vital Capacity (FVC) | 2 days
The change in Oxygen Saturation (SpO2) | 2 days
The change in Borg scale | 2 days
Device acceptance | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Ping-Hung Kuo, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Taiwan University Hospital, Taipei, Taiwan